CLINICAL TRIAL: NCT05178485
Title: Treatment Efficacy of Local Anesthetic/Steroid Mixture Injection for Patients With Odynophonia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Halted prematurely prior to enrollment of first participant
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ted Mau, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STU-2020-0443
Record Dates: First submitted 2021-12-08; First posted 2022-01-05 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Patients With a Diagnosis of Odynophonia
MeSH Terms: interventions — Bupivacaine; Triamcinolone; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled trial. A total of 40 subjects will be randomized to experimental group (receiving bupivacaine/triamcinolone mixture) or control group (receiving saline injection). Two injections will be given one week apart.
Who Masked: Care Provider, Investigator
Masking Description: Subjects will be blinded to group assignment. The physicians who are the treating providers of the subjects and who will perform the injections will also be blinded to group assignment. At each clinic visit for a subject's injection, the study coordinator will inform the clinic nurse of the group assignment, and the nurse will draw up the corresponding 2 mL injectate (either the bupivacaine/triamcinolone mixture or saline) and wrap the syringe in foil. The syringe will then be provided to the physician for the injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The experimental group (Experimental): At each clinic visit for a subject's injection, the study coordinator will inform the clinic nurse of the group assignment, and the nurse will draw up the corresponding 2 mL injectate (either the bupivacaine/triamcinolone mixture) and wrap the syringe in foil. The syringe will then be provided to the physician for the injection.
  Interventions: Drug: Bupivacain
- The control group (Placebo Comparator): At each clinic visit for a subject's injection, the study coordinator will inform the clinic nurse of the group assignment, and the nurse will draw up the corresponding 2 mL saline and wrap the syringe in foil. The syringe will then be provided to the physician for the injection.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Bupivacain — FDA approved drug
  Other Names: Kenalog-40
  Arms: The experimental group
Other: Normal Saline — FDA approved
  Arms: The control group

SUMMARY:
This is a double-blind, randomized, placebo-controlled trial. A total of 40 subjects will be randomized to experimental group (receiving bupivacaine/triamcinolone mixture) or control group (receiving saline injection). Two injections will be given one week apart. The primary outcome measure is the reduction in pain on the abbreviated McGill Pain Questionnaire (MPQ).

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled trial. A total of 40 subjects will be randomized to experimental group (receiving bupivacaine/triamcinolone mixture) or control group (receiving saline injection). Two injections will be given one week apart. The primary outcome measure is the reduction in pain on the abbreviated McGill Pain Questionnaire (MPQ).

The injection of a mixture of local anesthetic/steroid into the thyrohyoid membrane to target the internal branch of superior laryngeal nerve (SLN) has been shown to be effective for some patients with chronic cough. Although anecdotal experience suggests this injection may also be effective in alleviating neck pain in patients with odynophonia (pain associated with voicing), there are no prospective studies to define the efficacy of this injection for odynophonia. The purpose of the study is to conduct a randomized, placebo-controlled study on the effect of local anesthetic/steroid injection for patients with odynophonia.

Recruitment/Consent Patients with a diagnosis of odynophonia seen at the UT Southwestern Voice Center will be informed of the study and given the opportunity to participate. Consent will be carried out by the study team members.

Randomization Subjects will be assigned a Study ID sequentially by the study coordinator upon enrollment. Each study ID (from Subject 01 to Subject 40) will be a priori assigned to either the experimental group or the control group using a randomization function in Excel.

Blinding Subjects will be blinded to group assignment. The physicians who are the treating providers of the subjects and who will perform the injections will also be blinded to group assignment. At each clinic visit for a subject's injection, the study coordinator will inform the clinic nurse of the group assignment, and the nurse will draw up the corresponding 2 mL injectate (either the bupivacaine/triamcinolone mixture or saline) and wrap the syringe in foil. The syringe will then be provided to the physician for the injection.

Injections Injections will be performed in the usual fashion as for standard of care injections commonly performed. The subject will be seated in the exam chair with the chair slightly inclined to extend the neck.

Only unilateral injections will be performed even for patients with bilateral pain, so that the dose is the same for all subjects. Patients with bilateral pain will be asked to choose one side for the injection for the duration of the study. The patients will only be billed for a regular clinic visit and not for the actual injections.

Subjects in the Experimental Group will received a 2 mL injection consisting of 1 mL of 0.5% bupivacaine (5 mg bupivacaine-HCL) and 1 mL Kenalog-40 (40 mg triamcinolone acetonide). Subjects in the Control Group will receive 2 mL saline. A 1.5-in, 25G or 27G needle will be used.

Outcome Instruments The treatment progress/outcome will be based on questionnaires (modified version of McGill-Melzack Pain Questionnaire, Numeric Pain Scale, Brief Pain Inventory, Vocal Tract Discomfort scale and Voice Handicap Index-10) and the clinician's auditory-perceptual and acoustic analysis of voice. The data will be taken during the initial evaluation, at each treatment session, and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who report pain associated with voicing and are diagnosed with odynophonia

Exclusion Criteria:

* • Vocal fold mobility or tissue abnormality

  * history of jaw surgery/TMJ
  * history of neck surgery or trauma
  * Uncontrolled reflux. (patient's scoring on Reflux Symptom Index(RSI) is 13 or higher: Normative data suggests that a RSI of greater than or equal to 13 is clinically significant.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain on the McGill Pain Questionnaire | Baseline, Visit 2 (approximately 1 week)
  The McGill Pain Questionnaire (MPQ) is a valid and reliable measure of pain. The MPQ captures pain intensity on a 0 to 10 scale where 0 indicating no pain and 10 indicating severe pain

IPD SHARING:
Plan to Share IPD: No